CLINICAL TRIAL: NCT04577326
Title: A Single-Arm, Open-Label, Phase I Trial to Assess the Safety of Genetically Engineered Autologous T Cells Targeting the Cell Surface Antigen Mesothelin With Cell-Intrinsic Checkpoint Inhibition in Patients With Mesothelioma
Brief Title: Mesothelin-targeted CAR T-cell Therapy in Patients With Mesothelioma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Atara Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-328
Record Dates: First submitted 2020-09-30; First posted 2020-10-06 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Malignant Pleural Mesothelioma (MPM)
Keywords: Genetically Engineered Autologous T Cells; 20-328
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Cyclophosphamide; Immunotherapy, Adoptive

STUDY DESIGN:
Intervention Model Description: This is a phase I dose-escalation trial.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Engineered Autologous T Cells (Experimental): Following eligibility screening and enrollment, patients will undergo leukapheresis for the collection of peripheral blood mononuclear cells (PBMCs), to enable generation of M28z1XXPD1DNR. Following successful M28z1XXPD1DNR CAR T-cell manufacturing, patients will be reevaluated for eligibility. A preconditioning regimen of one dose of intravenous (IV) cyclophosphamide 1.5 g/m2 will be administered 2-7 days before the infusion. A single dose of M28z1XXPD1DNR CAR T cells will be instilled into the pleural cavity via a pleural catheter or through an interventional radiology-guided needle. All patients will be monitored in the hospital for a minimum of 48 h following the administration of CAR T cells.
  Interventions: Drug: cyclophosphamide; Biological: CAR T cells

INTERVENTIONS:
Drug: cyclophosphamide — A preconditioning regimen of one dose of intravenous (IV) cyclophosphamide 1.5 g/m^2 will be administered 2-7 days before the infusion.
Biological: CAR T cells — A single dose of M28z1XXPD1DNR CAR T cells will be instilled into the pleural cavity via a pleural catheter or through an interventional radiology-guided needle. Cohorts of 3 patients will be treated at each dose level, up to a maximum of 3 x 10^7 T cells/kg or until the MTD has been reached.

SUMMARY:
This study will test the safety of MSLN-targeted CAR-T cells at different doses to find the safest dose to give to people with MPM. The researchers want to see what effects, if any, the study treatment has on people with this type of cancer. This study is the first time that an MSLN-targeted CAR-T cell treatment with an anti-PD1 component is being given to people.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years
2. Karnofsky performance status ≥70%
3. Pathologically confirmed MPM

   1. Epithelioid or biphasic histologic diagnosis provided that ≥10% of the tumor expresses MSLN by IHC analysis
   2. Patients with peritoneal mesothelioma with pleural involvement are eligible only if there is radiographic and pathologic confirmation of mesothelioma in the pleural cavity and ≥10% of the tumor expresses MSLN by IHC analysis.
4. Previously treated with at least 1 treatment regimen
5. Measurable or evaluable disease (disease is considered evaluable but not measurable if it does not meet the eligibility criteria for mRECIST but is a manifestation of malignancy that can be followed qualitatively as an indicator of disease progression or treatment response)
6. Chemotherapy, targeted therapy, or radiotherapy must be completed at least 7 days before leukapheresis.

   a. CPI must be completed at least 21 days before leukapheresis.
7. Chemotherapy, targeted therapy, or therapeutic radiotherapy must be completed at least 14 days before administration of T cells.

   1. Palliative radiotherapy can be completed 2 days before lymphodepletion. Immunotherapy with CPI must be completed at least 42 days before administration of T cells.

9. Any major thoracic (thoracotomy with lung or esophageal resection) or abdominal (laparotomy with organ resection) operation must have occurred at least 28 days before study enrollment. Patients who have undergone diagnostic VATS or laparoscopy can be included in the study.

10. All acute toxic effects of any previous therapeutic or palliative radiotherapy, chemotherapy, or surgical procedures must have resolved to grade 1 (CTCAE v5.0).

11. Lab requirements (hematology):

a. Absolute neutrophil count ≥1.5 K/mcL b. Platelet count ≥100 K/mcL

12. Lab requirements (serum chemistry):

a. Bilirubin ≤1.5x upper limit of normal (ULN) b. Serum alanine aminotransferase and serum aspartate aminotransferase (ALT/AST) level ≤5x ULN c. Serum creatinine level ≤1.5x ULN or creatinine >1.5x ULN but calculated clearances of >60 by Cockcroft-Gault Equation

13. Negative screen for infectious disease markers including Hepatitis B core antibody, Hepatitis B surface antigen, Hepatitis C antibody, HIV 1-2 antibody, HTLV 1-2 and Syphilis (rapid plasma regain profile) Note - Patients with history of prior hepatitis B virus (HBV) infection are eligible if the HBV viral load is undetectable. Patients with a history of hepatitis C virus (HCV) infection who were treated for hepatitis C and cured are eligible if hepatitis C viral load is undetectable.

14. Life expectancy at the time of screening ≥4 months

Exclusion Criteria:

1. Patients receiving therapy for concurrent active malignancy

   a. Patients receiving treatment for in situ skin malignancies are not excluded.
2. Patients who received prior CAR T-cell therapy
3. Untreated or active central nervous system (CNS) metastases (progressing or requiring anticonvulsants or corticosteroids for symptomatic control). Patients with a history of treated CNS metastases are eligible if all the following criteria are met:

   1. Presence of measurable or evaluable disease outside of the CNS
   2. Radiographic demonstration of improvement upon completion of CNS-directed therapy and no evidence of interim progression between completion of CNSdirected therapy and the screening radiographic study
   3. Completion of radiotherapy ≥8 weeks before the screening radiographic study
   4. Discontinuation of corticosteroids and anticonvulsants ≥4 weeks before the screening radiographic study
4. History of seizure disorder
5. Active autoimmune disease that has required systemic treatment in the past year (with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs)

   a. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
6. Patients who are receiving daily systemic corticosteroids that are above physiological doses for any reason or who are under immunosuppressive or immunomodulatory treatment
7. Patients with the below cardiac conditions:

   1. New York Heart Association stage III or IV congestive heart failure
   2. Myocardial infarction ≤6 months before enrollment
   3. History of myocarditis
   4. Serious uncontrolled cardiac arrhythmia, unstable angina, or uncontrolled infection
8. Patients with left ventricular ejection fraction ≤40%
9. Patients with active interstitial lung disease/pneumonitis or a history of interstitial lung disease/pneumonitis requiring treatment with systemic steroids
10. Baseline pulse oximetry <90% on room air at the screening timepoint
11. Pregnant or lactating women

    a. Subjects and their partners with reproductive potential must agree to use an effective form of contraception during treatment and for 1 year following treatment.
12. Known active infection requiring antibiotic treatment 7 days before the start of treatment (Day 0). Note: treatment can be delayed at the discretion of the treating physician to allow the patient to recover from the infection.
13. Administration of live, attenuated vaccine within 8 weeks before the start of treatment (Day 0) and for 100 days following treatment.
14. Any other medical condition that, in the opinion of the PI, may interfere with a subject's participation in or compliance with the study
15. Any patient deemed to be noncompliant by the study team for administration of a high risk treatment agent and for close follow-up after treatment as required by the protocol
16. Patients with known hematologic malignancy requiring treatment in the preceding 5 years or a known history of lymphoid malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
MTD of M28z1XXPD1DNR | 2 years
  CTCAE v5.0 will be used to assess the severity of all treatment emerging toxicities/adverse events regardless

SECONDARY OUTCOMES:
overall response rate (ORR) | 2 years
  modified RECIST (mRECIST; v1.0)

CONTACTS AND LOCATIONS:
Overall Officials: Roisin O'Cearbhaill, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm